CLINICAL TRIAL: NCT02132364
Title: Controlled Education Of Patients After Stroke
Acronym: CEOPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011_34; 2012-A00473-40 (Other: ID-RCB number, ANSM); PHRIP 2012 - N°12-019-0306 (Other: DGOS)
Record Dates: First submitted 2014-05-05; First posted 2014-05-07 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2023-02

CONDITIONS: Stroke; Hypertension
Keywords: stroke; hypertension; secondary prevention; educational program
MeSH Terms: conditions — Stroke; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- optimised follow-up (Other): optimised follow-up will be done by nursing personnel associated with a caregiving member of his social circle.
  Interventions: Other: optimised follow-up
- typical follow-up (No Intervention): no intervention

INTERVENTIONS:
Other: optimised follow-up — optimised follow-up will be done by nursing personnel associated with a caregiving member of his social circle.
  Arms: optimised follow-up

SUMMARY:
The main objective of the study is to compare the benefit of optimised follow-up by nursing personnel from the vascular neurology department, including therapeutic follow-up and an educational program directed to the patient and a caregiving member of his social circle, with that of a typical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 60 years of age
* Patients who have had a first stroke, transient or permanent, ischaemic or haemorrhagic, justifying hospitalisation
* Patients with high blood pressure already treated or discovered at the time of the stroke and justifying the start of a treatment
* Patients who have had a stroke with sequelae allowing immediate return home or justifying a stay of less than one month in rehabilitation
* Patient having a member of his social circle who has agreed to provide follow-up for two years in association with the assigned nursing personnel in case of randomisation into the "optimised follow-up" group.

Exclusion criteria

* Patients less than 60 years of age
* Patients with a history of stroke
* Patients who do not have high blood pressure discovered by a treatment prior to the stroke or by abnormal blood pressure figures during hospitalisation
* Patients who have had a stroke causing serious sequelae, justifying an extended stay in a rehabilitation department
* Patient who has no one in his social circle capable of working with the assigned nursing personnel, or patient living in an institution

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2021-12-16 (Actual); Study Completion 2021-12-16 (Actual)

PRIMARY OUTCOMES:
blood pressure | 12 months
  blood pressure will be measured by nursing personnel who do not know the group into which the patient has been randomised.

SECONDARY OUTCOMES:
Outcome of stroke | 6 months 12 months 2 years.
  functional handicap (Rankin scale) cognitive state (MoCA scale)

CONTACTS AND LOCATIONS:
Overall Officials: REGIS BORDET, MD phD, Principal Investigator — University Hospital
Locations (17):
- France (17):
  - Chu Amiens Picardie, Amiens
  - CHU, Besançon
  - CHU, Bordeaux
  - Chru Brest, Brest
  - Hopital Pierre Wertheimer - Hcl, Bron
  - CH, Calais
  - Samsah Ghicl Capinghem, Capinghem
  - Ch Intercommunal Compiègne-Noyon - Compiegne, Compiègne
  - CHU, Dijon
  - Chu de Grenoble Alpes - Grenoble 9, Grenoble
  - CHRU, Lille
  - C H U Dupuytren Limoges, Limoges
  - Ch Sambre Avesnois Maubeuge, Maubeuge
  - Ch Saint Joseph, Paris
  - Chu La Miletrie - Poitiers, Poitiers
  - CHU, Rouen
  - Chru Nancy - Hopitaux de Braboi, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mendyk AM, Duhamel A, Bejot Y, Leys D, Derex L, Dereeper O, Detante O, Garcia PY, Godefroy O, Montoro FM, Neau JP, Richard S, Rosolacci T, Sibon I, Sablot D, Timsit S, Zuber M, Cordonnier C, Bordet R; on the behalf of Strokavenir network. Controlled Education of patients after Stroke (CEOPS)- nurse-led multimodal and long-term interventional program involving a patient's caregiver to optimize secondary prevention of stroke: study protocol for a randomized controlled trial. Trials. 2018 Feb 22;19(1):137. doi: 10.1186/s13063-018-2483-0. PMID 29471839
- [Derived] Crocker TF, Brown L, Lam N, Wray F, Knapp P, Forster A. Information provision for stroke survivors and their carers. Cochrane Database Syst Rev. 2021 Nov 23;11(11):CD001919. doi: 10.1002/14651858.CD001919.pub4. PMID 34813082